CLINICAL TRIAL: NCT07091318
Title: CBTi for the Treatment of Insomnia in Type 1 Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0987
Record Dates: First submitted 2025-04-24; First posted 2025-07-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 1; Insomnia
Keywords: insomnia; diabetes; sleep; adults; type 1 diabetes; stress; A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Initiation and Maintenance Disorders; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the treatment group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy Intervention for Insomnia (Experimental): Virtual CBTi sessions will be tailored to be address the specific challenges that come with type 1 diabetes.
  Interventions: Behavioral: Sleep quality improvement therapy
- Healthy Living (Active Comparator): Psychoeducation about general health and sleep alongside brief calls from a coach will be provided.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Sleep quality improvement therapy — 8 virtual CBTi sessions will be provided through a therapist weekly for the first four weeks and every other week for the last eight weeks of the study.
  Arms: Cognitive Behavioral Therapy Intervention for Insomnia
Behavioral: Healthy Living — Health education emails and brief coaching calls will be provided weekly. The phone coaches will not provide counseling or goal setting but can clarify what participants had questions on like terms and concepts.
  Arms: Healthy Living

SUMMARY:
The goal of this study is to learn if treating insomnia with a therapy intervention in people with type 1 diabetes will help to better control sugar levels, sleep, and quality of life. The questions this study aims to answer include:

Will this intervention help the insomnia symptoms? Will obtaining better sleep aid in the control of diabetes through measures like sugar levels? Will the intervention help with quality of life factors like mood and fatigue?

Researchers will compare participants receiving the therapy intervention for sleep with those in the "healthy living" intervention to see if the outcomes are different based on the treatment.

Participants in the therapy intervention group will:

* meet virtually with a therapist for 8 sessions via Zoom. Once a week for the first 4 weeks and then every other week for the last 4 sessions.

Participants in the healthy living group will:

* receive weekly health education emails
* receive brief weekly calls from a coach to answer any questions

Participants, regardless of intervention, over the 12 week study period will:

* monitor their sleep for 2 weeks through a sleep-monitoring watch
* share their continuous glucose monitoring data throughout the study
* answer questionnaires prior to the intervention, halfway through the intervention and then after the intervention
* attend 3 in person office visits

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 65 years old
* Have been diagnosed with Type 1 Diabetes for at least a year
* Use a continuous glucose monitor
* Have poor sleep quality
* Able to attend 3 office visits

Exclusion Criteria:

* Currently or planning pregnancy or breast feeding
* Employed with a rotating or night shift
* Are at a high risk for obstructive sleep apnea
* Non-English speaking (unable to participate in therapy or questionnaire).
* Take medications for sleep
* moderately severe to severe depression
* Have a significant medical history that includes conditions like heart failure, cirrhosis, COPD, diseases requiring oxygen, active treatment for cancer or psychiatric problems, history of stroke with neurological deficits, cognitive impairment, kidney failure that requires dialysis, illicit drug use, use of ADHD stimulant medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | From enrollment to the end of the intervention (12 weeks)
  Will be measured via the Acceptability of Intervention Measure (AIM) at the end of the interventions. AIM is measured through 4 questions on a scale of 1-5 resulting in scores from 4 to 20 points. The higher the score the higher the acceptability.

SECONDARY OUTCOMES:
Glycemic Variability | Week 0 (Baseline), 6 weeks (midpoint0 and 12 weeks (end of treatment)
  Assessed as time in, above or below range as collected by the continuous glucose monitor.
Pittsburgh Sleep Quality Index (PSQI) | Week 0 (baseline), Week 6 (midpoint) and Week 12 (end of treatment)
  The PSQI is a questionnaire that assesses sleep quality and disturbances within the last month. It consists of 18 questions that either have scaled questions with four options or asks the participant for input regarding factors like bed time, time to fall asleep, hours of sleep etc. Each participant answer, both on the scale and on input, is assigned a score between 0 and 3. Thus, the score range goes from 0 to 54, with a higher score indicating worse sleep quality.
Glycemic Control | Week 0 (baseline) and Week 12 (end of treatment)
  Assessed through A1C
Sleep duration | Week 0 (baseline) and Week 12 (end of treatment)
  Measured by actigraphy watch
Patient-Reported Outcomes Measurement Information System (PROMIS) for Sleep Disturbance | Week 0 (baseline), Week 6 (midpoint) and Week 12 (end of treatment)
  The PROMIS questionnaire assesses self-reported sleep quality through the lens of depth and restoration. It contains 8 questions regarding the last 7 days and is scored on a scale of 1 to 5 for each question. The scores range from 8 to 40. A higher score indicates worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Access to individual data will be restricted to the principle investigator and authorized members of the research team-- who will be trained on data confidentiality and how to handle secure data.